CLINICAL TRIAL: NCT02446613
Title: A Single-centre, Follow-up Study to Investigate the Effect of GSK2245035 on Nasal Allergic Reactivity in Subjects Who Completed Treatment in Study TL7116958 in 2014
Brief Title: Follow-up Study to Investigate the Effect of GSK2245035 on Nasal Allergic Reactivity in Subjects Completing Treatment in Study TL7116958
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 204509
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Asthma and Rhinitis
Keywords: Allergic Rhinitis; Nasal allergen challenge; Allergic Asthma; Effect on Allergen Reactivity
MeSH Terms: conditions — Asthma; Rhinitis; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal allergen challenge (Other): Subjects do not receive study medication in this study 204509. Subjects who carried from study TL7116958 treatment group GSK2245035 will undergo NAC with pollen allergen extract.
  Interventions: Other: Pollen allergen extract

INTERVENTIONS:
Other: Pollen allergen extract — Pollen (tree, grass or ragweed) allergen extracts will be provided by the research unit and diluted as required in normal saline. The specific pollen allergen extract that will be used for the nasal allergen challenge will be selected according to each subject's individual allergic sensitivity demonstrated in the previous study, TL7116958. If possible, extracts remaining from this study in 2014 will be used, provided they have not reached their expiry date.

SUMMARY:
This study will evaluate the duration of effect of GSK2245035 on allergic reactivity by repeating a nasal allergen challenge (NAC) approximately one year after treatment in subjects from TL7116958. This is a single centre, single period study in subjects with respiratory allergy/allergies who completed the study TL7116958 in 2014 to investigate the long term effect of previous treatment with GSK2245035 compared with placebo on total nasal symptoms elicited by nasal allergen challenge. Subjects and staff will remain blinded to the treatment received in the TL7116958 study (GSK2245035 or placebo). The study will consist of a screening visit to assess eligibility criteria, a study period consisting of a single visit when the nasal allergen challenge will be performed, and follow up by phone or a clinic visit at the discretion of the investigator 4-7 days following the allergen challenge. Eligible subjects will participate in this study for approximately70 days total from screening to follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with allergic rhinitis who completed study TL7116958 in 2014.
* Healthy as determined by the investigator or medically qualified designee based on a brief physical examination.
* Males and non-pregnant females.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Unresolved respiratory tract infection (RTI) at the time of study visit 2 NAC. Investigator discretion will be used regarding RTIs that have resolved during the 4 weeks preceding study visit 2.
* Unresolved asthma exacerbation requiring hospitalization and/or treatment with oral steroids or high doses of inhaled steroids at the time of study visit 2 NAC.

Investigator discretion will be used regarding exacerbations that have resolved since screening visit.

* A change in medical history since completion of the study TLR7116958 that in the opinion of the investigator and GlaxoSmithKline (GSK) medical monitor may pose additional risk factors.
* Subjects with a history of treatment with allergen-specific immunotherapy since completion of the TL7116958 study; subjects that have taken an investigational drug that, in the opinion of the investigator or designee, would have an effect on the nasal allergen challenge
* Subjects using steroid treatment (nasal steroids, 4 weeks; oral steroids, 4 weeks; inhaled steroids, 4 weeks) for allergic rhinitis and/or asthma prior to study visit 2, nasal allergen challenge
* Subjects using antihistamines (nasal antihistamines, 48 hours; oral antihistamines 72 hours), decongestants (nasal decongestants, 24 hours; oral decongestants, 24 hours.), prior to study visit 2, nasal allergen challenge.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2015-08-10 (Actual); Study Completion 2015-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 204509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par) of All subjects population (ASP) from study TL7116958 who passed screening for study 204509 were used as safety population for this study. All outputs using information from study TL7116958 were analyzed using ASP and stand alone outputs for this study were analyzed using Safety population.
Pre-assignment Details: Participants with respiratory allergy/allergies, with or without asthma, who completed the parent study TL7116958 in 2014 were enrolled to investigate the long term effect of previous treatment with GSK2245035 compared to placebo on total nasal symptoms (sym.) elicited by allergen challenge.
Groups:
- Placebo Once Weekly: Participants were not administered with placebo during the current study (204509). Participants were subjected to nasal allergen challenge (NAC) at Visit 2 to investigate the long term effect of matching placebo, intranasal (i.n.), administered once weekly during the parent study (TL7116958). Total and individual nasal sym. were recorded up to 6 hours (h) post NAC.
- GSK2245035 20 ng, i.n., Once Weekly: Participants were not administered with study medication in the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of GSK2245035 20 nanograms (ng), i.n., once weekly received during the parent study (TL7116958). Total and individual nasal sym. were recorded up to 6 h post NAC.
Period: Overall Study
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Started | 6 | 10
Completed | 6 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Once Weekly: Participants were not administered with placebo during the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of matching placebo, i.n., administered once weekly during the parent study (TL7116958). Total and individual nasal sym. were recorded up to 6 h post-NAC.
- GSK2245035 20 ng, i.n., Once Weekly: Participants were not administered with study medication in the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of GSK2245035 20 ng, i.n., once weekly received during the parent study (TL7116958). Total and individual nasal sym. were recorded up to 6 h post-NAC.
- Total: Total of all reporting groups
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (12.82) | 40.4 (12.02) | 40.8 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 10 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Total Nasal Sym. Score (TNSS) at Post-NAC 15 Minutes (Min)
Description: TNSS was obtained from 4 individual nasal sym. including nasal congestion, rhinorrhoea, nasal itch and sneezing. Participants rated sym. on a 4-point scale. For nasal blockage and congestion the scores were (0= Breathing through nose freely and easily, 1= Slight difficulty breathing through nose, 2= Moderate difficulty breathing through nose and 3= Severe difficulty breathing through nose). For rhinorrhoea, nasal itching and sneezing (0= None: No sym. whatsoever; Absent, 1= Mild: Sym. is present, noticeable but not bothersome, 2= Moderate: Sym. is bothersome, but tolerable and 3= Severe: Sym. which are bothersome, harder to tolerate). The individual sym. scores were combined to produce a TNSS. TNSS were reported as median (credible interval). The baseline values were the latest pre-dose assessments. Change from baseline was measured as the value recorded at 15 min post-NAC minus Baseline value.
Time Frame: Day 1 (Baseline [pre-NAC] and post-NAC 15 min)
Population: The Safety population consisted of members of the ASP of parent study TL7116958 who had passed screening for study 204509.
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Score on a scale | 3.8 [1.22 to 6.53] | 5.9 [3.91 to 7.81]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-1.41 to 5.43], Standard Deviation 0.007 — The posterior probability statement value for change from baseline in post-challenge TNSS ≤0 was 0.1071

2. Primary Outcome: Mean Change From Baseline in the TNSS Over Post-NAC 1 h
Description: TNSS was obtained from 4 individual nasal sym. including nasal congestion, rhinorrhoea, nasal itch and sneezing. Participants rated sym. on a 4-point scale. For nasal blockage and congestion the scores were (0= Breathing through nose freely and easily, 1= Slight difficulty breathing through nose, 2= Moderate difficulty breathing through nose and 3= Severe difficulty breathing through nose). For rhinorrhoea, nasal itching and sneezing (0= None: No sym. whatsoever; Absent, 1= Mild: Sym. is present, noticeable but not bothersome, 2= Moderate: Sym. is bothersome, but tolerable and 3= Severe: Sym. which are bothersome, harder to tolerate). The individual sym scores were combined to produce a TNSS. TNSS were reported as median (credible interval). The baseline values were the latest pre-dose assessments. Change from baseline was measured as the value recorded at a specified time point minus Baseline value. Weighted mean (WM) 0-1h of 15, 30 min and 1 h was reported.
Time Frame: Day 1 (Baseline [pre-NAC], 15 to post-NAC 1h)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Score on a scale
Groups:
- GSK2245035 20 ng, i.n., Once Weekly: Participants were not administered with study medication in the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of GSK2245035 20 ng, i.n., once weekly received during the parent study (TL7116958) . Total and individual nasal sym. were recorded up to 6 h post-NAC.
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Score on a scale | 2.4 [0.24 to 4.63] | 3.4 [1.70 to 4.96]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.98 to 3.75], Standard Deviation 0.007 — The posterior probability statement value for change from baseline in post-challenge TNSS ≤0 was 0.2417

3. Primary Outcome: Mean Change From Baseline in the TNSS Over Post-NAC 6 h
Description: TNSS was obtained from 4 individual nasal sym. including nasal congestion, rhinorrhoea, nasal itch and sneezing. Participants rated sym. on a 4-point scale. For nasal blockage and congestion the scores were (0= Breathing through nose freely and easily, 1= Slight difficulty breathing through nose, 2= Moderate difficulty breathing through nose and 3= Severe difficulty breathing through nose). For rhinorrhoea, nasal itching and sneezing (0= None: No sym. whatsoever; Absent, 1= Mild: Sym. is present, noticeable but not bothersome, 2= Moderate: Sym. is bothersome, but tolerable and 3= Severe: Sym. which are bothersome, harder to tolerate). The individual sym scores were combined to produce a TNSS. TNSS were reported as median (credible interval). The baseline values were the latest pre-dose assessments. Change from baseline was measured as value recorded at a specified time point minus Baseline value. WM 0-6 h of 15, 30 min, 1, 2, 3, 4, 5, 6h was reported.
Time Frame: Day 1 (Baseline [pre-NAC] to post-NAC 6 h)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Score on a scale
Groups:
- GSK2245035 20 ng, i.n., Once Weekly: Participants were not administered with study medication in the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of GSK2245035 20 ng, i.n., once weekly received during the parent study (TL7116958). Total and individual nasal sym were recorded up to 6 h post-NAC.
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Score on a scale | 1.2 [0.04 to 2.33] | 1.6 [0.73 to 2.44]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Median Difference (Final Values) = 0.4, 95% CI 2-sided [-1.08 to 1.87], Standard Deviation 0.007 — The posterior probability statement value for change from baseline in post-challenge TNSS ≤0 was 0.2876

4. Primary Outcome: Maximum (Max) Mean Change From Baseline (BL) in the TNSS Over Post-NAC 6 h
Description: TNSS was obtained from 4 individual nasal sym.: nasal congestion, rhinorrhoea, nasal itch and sneezing. Par rated sym. on a 4-point scale. For nasal blockage and congestion the scores were (0= Breathing through nose freely and easily, 1= Slight difficulty breathing through nose, 2= Moderate difficulty breathing through nose and 3= Severe difficulty breathing through nose). For rhinorrhoea, nasal itching and sneezing (0= None: No sym. whatsoever; Absent, 1= Mild: Sym. is present, noticeable but not bothersome, 2= Moderate: Sym. is bothersome, but tolerable and 3= Severe: Sym. which are bothersome, harder to tolerate). The individual sym. scores were combined to produce a TNSS. TNSS were reported as median (credible interval). BL values were the latest pre-dose assessments. Change from BL was measured as the value recorded at a specified time point minus BL value. The max change from BL from the set of individual PNIF % reduction measurements made over the 0 to 6 h sampling period.
Time Frame: Day 1 (Baseline [pre-NAC] to post-NAC 6 h)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Score on a scale
Groups:
- Placebo Once Weekly: Participants were not administered with placebo during the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of matching placebo, i.n., administered once weekly during the parent study (TL7116958). Total and individual nasal sym were recorded up to 6 h post-NAC.
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Score on a scale | 4.1 [1.41 to 6.80] | 5.9 [3.83 to 7.87]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Median Difference (Final Values) = 1.9, 95% CI 2-sided [-1.86 to 5.34], Standard Deviation 0.006 — The posterior probability statement value for change from baseline in post-challenge TNSS ≤0 was 0.1453

5. Primary Outcome: Percent Change From Baseline in the Peak Nasal Inspiratory Flow (PNIF) at Post-NAC 15 Min
Description: PNIF data recorded at Baseline pre-challenge and at 15, 30 min and 1h. The percent change from Baseline and at specified time point was derived by the formula (PNIF at Baseline minus PNIF at Post-NAC specified time point) divided by PNIF at Baseline) multiplied by 100. The baseline values were the latest pre-dose assessments. The baseline value were the latest pre-dose assessments. Percent change in PNIF were reported as median (credible interval). WM 0-1 h of 15, 30 min and 1 h was reported. WM were derived by first calculating the AUC using the trapezoidal rule, and then dividing by the time interval. If available, actual times were used in the calculation, otherwise planned relative times were used for the calculation.
Time Frame: Day 1 (Baseline [pre-NAC] and post-NAC 15 min)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Percent change
Groups:
- GSK2245035 20 ng, i.n., Once Weekly: Participants were not administered with study medication in the current study (204509). Participants were subjected to NAC at Visit 2 to investigate the long term effect of GSK2245035 20 ng, i.n., once weekly received during the parent study (TL7116958) . Total and individual nasal sym were recorded up to 6 h post-NAC.
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Percent change | 27.6 [15.87 to 39.63] | 32.2 [23.71 to 40.72]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Median Difference (Final Values) = 4.6, 95% CI 2-sided [-10.70 to 19.71], Standard Deviation 0.006 — The posterior probability statement value for percentage reduction in the reductions of PNIF ≤0 was 0.2665

6. Primary Outcome: Percent Change From Baseline in the PNIF Over Post-NAC 1 h
Description: PNIF data recorded at Baseline pre-challenge and at 15, 30 min and 1h. The percent change from Baseline and at specified time point was derived by the formula (PNIF at Baseline minus PNIF at Post-NAC specified time point) divided by PNIF at Baseline) multiplied by 100. The baseline values were the latest pre-dose assessments. Percent change in PNIF were reported as median (credible interval). WM 0-1 h of 15, 30 min and 1 h was reported. WM were derived by first calculating the AUC using the trapezoidal rule, and then dividing by the time interval. If available, actual times were used in the calculation, otherwise planned relative times were used for the calculation.
Time Frame: Day 1 (Baseline [pre-NAC] to post-NAC 1 h)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Percent change | 20.8 [5.45 to 35.84] | 25.0 [14.69 to 36.05]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Median Difference (Final Values) = 4.3, 95% CI 2-sided [-14.97 to 24.38], Standard Deviation 0.007 — The posterior probability statement value for percentage reduction in the reductions of PNIF ≤0 was 0.3266

7. Primary Outcome: Percent Change From Baseline in the PNIF up to Post-NAC 6 h
Description: PNIF data recorded at Baseline pre-challenge and at 15, 30 min, 1, 2, 3, 4, 5, 6h. The percent change from Baseline and at specified time point was derived by the formula (PNIF at Baseline minus PNIF at Post-NAC specified time point) divided by PNIF at Baseline) multiplied by 100. The baseline values were the latest pre-dose assessments. Percent change in PNIF were reported as median (credible interval). WM 0-6h of 15, 30 min, 1, 2, 3, 4, 5, 6h was reported. WM were derived by first calculating the AUC using the trapezoidal rule, and then dividing by the time interval. If available, actual times were used in the calculation, otherwise planned relative times were used for the calculation.
Time Frame: Day 1 (Baseline [pre-NAC] to post-NAC 6 h)
Population: Safety populaton
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Percent change | 6.3 [-7.56 to 20.47] | 7.3 [-2.98 to 17.68]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Median Difference (Final Values) = 1.1, 95% CI 2-sided [-17.47 to 19.20], Standard Deviation 0.008 — The posterior probability statement value for percentage reduction in the reductions of PNIF ≤0 was 0.4528

8. Primary Outcome: Maximum Percent Change From Baseline in PINF Over Post-NAC 6 h
Description: PNIF data recorded at Baseline pre-challenge and at 15, 30 min, 1, 2, 3, 4, 5, 6h. The percent change from Baseline and at specified time point was derived by the formula (PNIF at Baseline minus PNIF at Post-NAC specified time point) divided by PNIF at Baseline) multiplied by 100. The baseline values were the latest pre-dose assessments. Percent change in PNIF were reported as median (credible interval). Maximum change from Baseline till 6h was reported.
Time Frame: Day 1 (Baseline [pre-NAC] to post-NAC 6 h)
Population: Safety population
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Percent change | 33.3 [16.89 to 49.33] | 39.9 [29.18 to 51.53]
Statistical Analysis 1: Comparison: Placebo Once Weekly vs GSK2245035 20 ng, i.n., Once Weekly; Test type: Superiority or Other; Median Difference (Final Values) = 6.6, 95% CI 2-sided [-13.69 to 28.04], Standard Deviation 0.007 — The posterior probability statement value for percentage reduction in the reductions of PNIF ≤0 was 0.2525

9. Secondary Outcome: Mean Change From Baseline in Individual Nasal Sym. Including Sneezing, Nasal Congestion, Rhinorrhoea and Nasal Itch.
Description: Four individual nasal sym. including nasal congestion, rhinorrhoea, nasal itch and sneezing were recorded at Baseline (pre-NAC) and at post-NAC 15, 30 min, 1, 2, 3, 4, 5, 6h. Participants rated sym. on a 4-point scale. For nasal blockage and congestion the scores were (0= Breathing through nose freely and easily, 1= Slight difficulty breathing through nose, 2= Moderate difficulty breathing through nose and 3= Severe difficulty breathing through nose). For rhinorrhoea, nasal itching and sneezing (0= None: No sym. whatsoever; Absent, 1= Mild: Sym. is present, noticeable but not bothersome, 2= Moderate: Sym. is bothersome, but tolerable and 3= Severe: Sym. which are bothersome, harder to tolerate). The baseline value were the latest pre-dose assessments. Mean change from Baseline at 15 min, WM0-1h, WM 0-6h, and maximum change over 0-6 h were reported. Change from Baseline was measured as the value recorded at a specified time point minus Baseline value.
Time Frame: Day 1 (Baseline [pre-NAC] to post-NAC 6 h)
Population: Safety population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Number analyzed (Participants) | 6 | 10
Score on a scale
  Sneezing, 15 min | 1.33 (1.366) | 1.50 (1.080)
  Sneezing, WM 0-1 h | 0.56 (0.706) | 0.56 (0.641)
  Sneezing, WM 0-6 h | 0.40 (0.496) | 0.19 (0.463)
  Sneezing, Max 0-6 h | 1.33 (1.366) | 1.60 (1.075)
  Rhinorrhoea, 15 min | 0.50 (0.548) | 1.60 (1.075)
  Rhinorrhoea, WM 0-1 h | 0.15 (0.300) | 1.16 (0.924)
  Rhinorrhoea, WM 0-6 h | -0.06 (0.383) | 0.60 (0.791)
  Rhinorrhoea, Max 0-6 h | 0.50 (0.548) | 1.60 (1.075)
  Nasal itching , 15 min | 0.67 (1.033) | 1.50 (0.850)
  Nasal itching , WM 0-1 h | 0.44 (0.832) | 1.15 (0.733)
  Nasal itching , WM 0-6 h | 0.05 (0.684) | 0.60 (0.556)
  Nasal itching , Max 0-6 h | 0.83 (0.753) | 1.60 (0.843)
  Nasal blockage , 15 min | 1.17 (0.753) | 1.70 (0.675)
  Nasal blockage , WM 0-1 h | 0.73 (0.533) | 1.26 (0.641)
  Nasal blockage , WM 0-6 h | 0.43 (0.485) | 0.64 (0.500)
  Nasal blockage , Max 0-6 h | 1.33 (0.816) | 1.80 (0.632)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from participant's consent for participation in the study till follow-up contact (4 to 7 day post Visit 2). Adverse events (AEs) were collected from the start of Study Visit 2 NAC until the follow-up contact.
Description: Safety population was used to record AEs and SAEs. No SAEs were reported in the study.
Arm/Group | Placebo Once Weekly | GSK2245035 20 ng, i.n., Once Weekly
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Once Weekly (N=6) | GSK2245035 20 ng, i.n., Once Weekly (N=10)
Urinary tract infection (Infections and infestations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.